CLINICAL TRIAL: NCT02025439
Title: Amantadine + rTMS as a Neurotherapeutic for Disordered Consciousness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edward Hines Jr. VA Hospital (U.S. Federal Agency)
Responsible Party: Principal Investigator, Theresa Pape, Clinical Neuroscientist, Edward Hines Jr. VA Hospital
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1R21HD075192 (NIH)
Record Dates: First submitted 2013-12-23; First posted 2014-01-01 (Estimated); Results first posted 2020-08-24 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury; Transcranial Magnetic Stimulation; Amantadine; Vegetative State; Minimally Conscious State
MeSH Terms: conditions — Brain Injuries, Traumatic; Persistent Vegetative State | interventions — Transcranial Magnetic Stimulation; Amantadine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rTMS Alone followed by rTMS+AMA (Experimental): Subjects assigned to rTMS Alone will receive 30 sessions of rTMS. Two rTMS sessions will be provided per day, four days per week.After first completing rTMS Alone, subjects will receive rTMS plus Amantadine. A total of 30 rTMS sessions are provided, 2 rTMS sessions per day, four days per week, while receiving 200mg of Amantadine daily.
  Interventions: Device: rTMS; Drug: Amantadine
- AMA Alone followed by rTMS+AMA (Experimental): Subjects who are assigned to the Amantadine Alone group will receive 28 doses of Amantadine (100mg BID) every day for 28 days. After first completing Amantadine Alone subjects will receive rTMS plus Amantadine. A total of 30 rTMS sessions are provided, 2 rTMS sessions per day, four days per week, while receiving 200mg of Amantadine daily.
  Interventions: Device: rTMS; Drug: Amantadine

INTERVENTIONS:
Device: rTMS
  Other Names: Repetitive Transcranial Magnetic Stimulation
Drug: Amantadine
  Other Names: Symadine; Symmetrel

SUMMARY:
The purpose of this study is to examine the safety and efficacy of repetitive transcranial magnetic stimulation (rTMS) combined with Amantadine relative to rTMS Alone and Amantadine Alone for persons in chronic states of seriously impaired consciousness. The hypothesis is that provision of rTMS+Amantadine will provide a safe yet synergistic effect that induces or accelerates functional recovery.

DETAILED DESCRIPTION:
The R21 research objective is to examine the safety and efficacy of repetitive transcranial magnetic stimulation (rTMS) combined with Amantadine (TMS + Amantadine) relative to rTMS Alone and Amantadine Alone for persons in chronic states of seriously impaired consciousness. The hypothesis is that provision of rTMS+Amantadine will provide a safe yet synergistic effect that induces or accelerates functional recovery. This hypothesis is based on (a) preliminary data indicating partially improved neurobehavioral functioning mechanistically related to rTMS-induced neural activity and connectivity as well as improved integrity of white fiber tracts, (b) relationship between dopamine (DA) and common traumatic brain injury (TBI) impairments, (c) role of DA in mediating consciousness, (d) the commonality between and DA and rTMS-targeted pathways, (e) clinical efficacy and safety of Amantadine, (f) mechanisms of action of Amantadine, and (g) the association between rTMS and Amantadine with up-regulating brain derived neurotrophic factor. The rationale is that pairing rTMS with Amantadine will have a complementary and synergistic effect on factors promoting conscious behavior. The specific aims are to: (1) Demonstrate that rTMS+Amantadine is safely tolerated, (2) Determine neurobehavioral effect of rTMS+Amantadine, and (3) Characterize pre-and post-treatment neural changes in neural activation. Aim 1 is based on our preliminary safety data and safety data regarding Amantadine. To address Aims 2 & 3 we use a repeated measures baseline control design with randomized treatment orders yielding three treatment groups; rTMS + Amantadine, rTMS Alone and Amantadine Alone. Analyses for Aims 2 and 3 involve comparing these treatment groups according to neurobehavioral growth trajectories, mean amount of neural activation and connectivity within and between brain regions, and indices of fiber tract directionality.

ELIGIBILITY:
Inclusion Criteria:

* 18-64 years of age
* Suffered a severe brain injury of traumatic origin at least 1-year prior to study enrollment
* Remain in a state of disordered consciousness
* Brain injuries will include injury with resulting coup-contre-coup injuries, excluding persons with trauma due to blunt injuries and/or non-traumatic encephalopathy

Exclusion Criteria:

* Have 1 or more Amantadine contraindications: On monoamino oxidase inhibitor-B, hypersensitivity/idiosyncrasy to sympathomimetic amines, uncontrolled hypertension, glaucoma or Congestive Heart Failure
* Have contraindications to Amantadine Dose of 200 mg Daily as determined by estimated Glomerular Filtration Rate (eGFR) ≤ 60 (ml/min)
* Abnormal results of Liver Function Test at screening
* Receiving anti-epileptic medications to control active seizures or have had a documented seizure within three months of study enrollment
* Incurred large cortically based ischemic infarction/encephalomalacia subsequent to TBI
* Have documented history of previous TBI, psychiatric illness (DSM criteria) and/or organic brain syndrome such as Alzheimer's
* Are using medications which may interfere with Amantadine and cannot be safely titrated or discontinued
* Are pregnant
* Have implanted cardiac pacemaker or defibrillator, cochlear implant, nerve stimulator, intracranial metal clips
* Have MRI and/or TMS contraindications such as: History of claustrophobia, metal in eyes/face, shrapnel/bullet remnants in brain
* Are fully conscious as indicated by a score of 6 on the Motor Function scale and/or a score of 2 on the Communication scale of the CRS-R,
* Are within first year of injury
* Are <18 years of age and > 65 years of age
* Have an injury or condition due to blunt trauma only or non-traumatic encephalopathy
* Have programmable CSF shunt or are ventilator dependent

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2014-02; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theresa BenderPape, DrPH, Principal Investigator — Edward Hines Jr. VA Hospital
Locations (2):
- United States (2):
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Edward Hines, Jr. VA Hospital, Hines, Illinois

REFERENCES:
- [Background] Pape TL, Rosenow J, Lewis G. Transcranial magnetic stimulation: a possible treatment for TBI. J Head Trauma Rehabil. 2006 Sep-Oct;21(5):437-51. doi: 10.1097/00001199-200609000-00063. PMID 16983227
- [Background] Louise-Bender Pape T, Rosenow J, Lewis G, Ahmed G, Walker M, Guernon A, Roth H, Patil V. Repetitive transcranial magnetic stimulation-associated neurobehavioral gains during coma recovery. Brain Stimul. 2009 Jan;2(1):22-35. doi: 10.1016/j.brs.2008.09.004. Epub 2008 Oct 23. PMID 20633400

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: nothing to report
Groups:
- rTMS Alone Followed by rTMS+AMA: Subjects assigned to rTMS Alone will receive 30 sessions of rTMS. Two rTMS sessions will be provided per day, four days per week.upon completion of assigned treatment order, the subject will then receive 30 sessions of combination therapy of rTMS + Amantadine
  rTMS
- AMA Alone Followed by rTMS+AMA: Subjects who are assigned to the Amantadine Alone group will receive 28 doses of Amantadine (100mg BID) every day for 28 days. upon completion of assigned treatment order, the subject will then receive 30 sessions of combination therapy of rTMS + Amantadine
  Amantadine
Period: Overall Study
Arm/Group | rTMS Alone Followed by rTMS+AMA | AMA Alone Followed by rTMS+AMA
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- rTMS First: Subjects assigned to rTMS Alone will receive 30 sessions of rTMS. Two rTMS sessions will be provided per day, four days per week.
  rTMS
- Amantadine First: Subjects who are assigned to the Amantadine Alone group will receive 28 doses of Amantadine (100mg BID) every day for 28 days.
  Amantadine
- Total: Total of all reporting groups
Arm/Group | rTMS First | Amantadine First | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 24 [21 to 27] | 33 [28 to 37] | 28 [21 to 37]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Intensity of Adverse Event
Description: If an adverse event occurred, the intensity was also indicated. The intensity of an adverse event was determined using a scale from 1-5 with 5 being the worst. The purpose of the study is to examine safety of rTMS combined with AMA relative to rTMS Alone and AMA alone. Results are not reported "per arm" rather, the arms are combined so as to compare the outcome when the interventions are provided separately (i.e., rTMS alone and amantadine alone) vs interventions are combined (rTMS +Amantadine alone).
Time Frame: 30 days after treatment "alone" and an additional 30 days after treatment "combined" (i.e., 60 days)
Population: Results are reported both "per arm" at the end of 30 days when a single treatment (either rTMS or AMA) was ended, and additional results are reported with both arms combined to report the outcome after 60 days
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- rTMS Alone: Subjects assigned to start with rTMS Alone
- rTMS+AMA: All subjects that received rTMS plus Amantadine. A total of 30 rTMS sessions are provided, 2 rTMS sessions per day, four days per week, while receiving 200mg of Amantadine daily.
- AMA Alone: Subjects assigned to start with amantadine alone
Arm/Group | rTMS Alone | rTMS+AMA | AMA Alone
Number analyzed (Participants) | 2 | 4 | 2
score on a scale | 0.5 (0.52) | 0.98 (0.38) | 0.33 (0.51)
Statistical Analysis 1: Comparison: rTMS Alone vs rTMS+AMA; Test type: Other; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 0.071

ADVERSE EVENTS:
Time Frame: 3 months and 6 months
Description: A Clinical Data Monitoring Log was used to record. Most were collected daily. CNS changes were collected once during MRI scan. clinical indices include fatigue, fever, hypertension, hypotension, infection at IV site, weight loss/gain, seizures, skin breakdown at IV site, skin breakdown on scalp, general skin breakdown, sweating and neurochecks hourly between rTMS sessions on the same day.
Groups:
- rTMS Alone: Subjects assigned to rTMS Alone 30 sessions of rTMS. Two rTMS sessions will be provided per day, four days per week.
- rTMS+AMA: Subjects who are assigned to the Amantadine Alone group will receive 28 doses of Amantadine (100mg BID) every day for 28 days.Then, A total of 30 rTMS sessions are provided, 2 rTMS sessions per day, four days per week, while receiving 200mg of Amantadine daily.
- AMA Alone: Subjects who are assigned to the Amantadine Alone group will receive 28 doses of Amantadine (100mg BID) every day for 28 days.
Arm/Group | rTMS Alone | rTMS+AMA | AMA Alone
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/4 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/4 | 0/2
Other Adverse Events (participants affected / at risk) | 2/2 | 4/4 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rTMS Alone (N=2) | rTMS+AMA (N=4) | AMA Alone (N=2)
Fatigue (General disorders) | 2 (2) | 2 (19) | 1 (4)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0)
hypertension (General disorders) | 1 (1) | 2 (7) | 0 (0)
Hypotension (General disorders) | 0 (0) | 2 (10) | 1 (8)
Infection at IV site (General disorders) | 0 (0) | 2 (2) | 0 (0)
Weight Loss (General disorders) | 0 (0) | 1 (2) | 0 (0)
Neurocheck (General disorders) | 2 (3) | 3 (8) | 0 (0)
Seizure (General disorders) | 0 (0) | 0 (0) | 0 (0)
Skin breakdown at venous site (General disorders) | 0 (0) | 1 (4) | 0 (0)
General Skin Integrity (General disorders) | 0 (0) | 1 (2) | 0 (0)
Skin breakdown at scalp (General disorders) | 0 (0) | 1 (4) | 0 (0)
Sweating (General disorders) | 1 (1) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No